CLINICAL TRIAL: NCT07037121
Title: Healthy Eating Adherence & Routine Transformation Through a Kitchen Makeover Whole-Food, Plant-Based Diet Jumpstart (HEARTKITCHEN)
Brief Title: HEART Kitchen Pilot
Acronym: HEARTKITCHEN
Status: Withdrawn | Phase: Not Applicable | Type: Interventional
Why Stopped: PI leaving
Sponsor: Reya Andrews (Other)
Responsible Party: Sponsor-Investigator, Reya Andrews, Principal Investigator, University of Kentucky
Organization: University of Kentucky (Other)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 100837
Record Dates: First submitted 2025-06-16; First posted 2025-06-25 (Actual); Last update posted 2025-08-11 (Actual); Status verified 2025-08

CONDITIONS: Cardiovascular Diseases; Type 2 Diabetes; Obesity and Obesity-related Medical Conditions
Keywords: Whole-Food Plant-Based Diet; Cardiovascular Disease; Health Disparities; Feasibility Study; Public Housing; Spousal Support; Low-Income Adults; Diet Adherence; Nutrition Intervention; Kitchen Makeover
MeSH Terms: conditions — Cardiovascular Diseases; Diabetes Mellitus, Type 2; Obesity

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Whole Food Plant Based (WFPB) Diet (Experimental): 28 day kitchen makeover to include initial grocery supplies, cooking equipment, recipes, and meal-prep instruction, and nutrition counseling by a licensed nutritionist, and educational support materials
  Interventions: Behavioral: Whole Food Plant Based Diet Jumpstart

INTERVENTIONS:
Behavioral: Whole Food Plant Based Diet Jumpstart — Participants receive personally-tailored support by a research nutritionist during five total visits: (1)baseline visit to collect surveys on health status, current home kitchen-based habits, kitchen inventory, food preferences, and clinical measures, followed by assessing health goals, obstacles, and opportunities. At least two breakfast, three lunch, and five dinner WFPB recipes will be selected. (2) A kitchen-centered visit will target the fridge, pantries, and cabinets to assist participants in cleaning out ultra-processed "junk" foods. These foods will be stored in a large tote during the study. (3) The day before the intervention starts will be a grocery shopping trip to purchase the WFPB heart-healthy groceries together. (4) Intervention day 1 will focus on jumpstarting meal prep. After day 1, weekly 30-min telehealth nutrition consultations will provide additional support. (5) Clinical measures and postintervention surveys will be collected on day 29.

SUMMARY:
This study is testing a 28-day healthy eating program for adults who live in public housing and are at risk for heart disease. The program helps people eat more whole plant foods, like fruits, vegetables, beans, and whole grains, and avoid foods that are highly processed or high in fat. Participants get a "kitchen makeover," including groceries, cooking tools, whole-food, plant-based recipes, and support from a nutritionist. The goal is to see if the program is easy to follow, helpful, and if support from a spouse or partner makes it easier to stick with the new way of eating.

The study will include 24 adults who either have heart disease or are at risk because of conditions like high blood pressure, diabetes, or obesity. Researchers will visit participants at home to provide supplies and support. They will also collect surveys, interviews, and health information to learn more about how the program worked and how well participants followed the diet.

ELIGIBILITY:
Inclusion Criteria:

* Adult public housing residents who have been diagnosed with cardiovascular disease (Individuals who have had a documented history of myocardial infarction; Individuals who have ever had a positive stress test;, Individuals who have undergone coronary artery bypass grafting surgery at any point in their life)
* meet at least 2 of the criteria for metabolic syndrome: abdominal obesity (waist circumference of more than 35 inches for women and more than 40 inches for men or BMI = 30), high triglycerides (>150 mg/dL or drug treatment for elevated TG), low HDL cholesterol (<40 mg/dL for men and < 50 mg/dL for women or drug treatment for reduced HDL-C), high blood pressure (=130 mm Hg systolic BP, =85 mm Hg diastolic BP, or drug treatment for hypertension), high fasting blood glucose (> or = 100 mg/dL or drug treatment for elevated glucose or prediabetes/ type 2 diabetes diagnosis)
* able to provide written informed consent
* fluent in the English language

Exclusion Criteria:

* Active cancer or chronic kidney disease diagnosis or are undergoing cancer or dialysis treatment
* any food allergies or dietary restrictions that would prevent them from adhering to a whole-food, plant-based (WFPB) diet
* an existing or former neurological disorder or a neuropsychiatric disorder that affects decision-making ability
* current smoking
* current excessive alcohol intake
* recent history of drug abuse
* morbid obesity (BMI > 40)
* history of bariatric surgery
* pregnant or lactating
* current use of a WFPB (excludes all animal-based foods) or vegan diet

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2025-09 (Estimated); Primary Completion 2025-11 (Estimated); Study Completion 2025-11 (Estimated)

PRIMARY OUTCOMES:
Change in adherence to the whole-food, plant-based (WFPB) diet (pre-post) based on ACLM diet screener. | Baseline and post intervention (week 4)
  Dietary intake will be assessed using the American College of Lifestyle Medicine (ACLM) Diet Screener at baseline (Day 0) and post-intervention (Day 29). This validated 15-item tool measures frequency of consumption of foods consistent with a whole-food, plant-based (WFPB) diet. Total scores range from 0 to 100, with higher scores indicating greater adherence to a WFPB diet. Change in dietary intake will be calculated by subtracting the baseline score from the post-intervention score. Positive values reflect improvement in WFPB dietary adherence.
Change in weight | Baseline and week 4
  Weightwill be measured using the Runstar Scale for Body Weight and Fat Percentage, 8 Electrodes High Precision Digital Scale
Change in Body Mass Index | Baseline and week 4
  BMI in kg/m^2 based on measured weight in kg and height in meters.
Change in fat mass | Baseline and week 4
  Fat mass will be measured using the Runstar Scale for Body Weight and Fat Percentage, 8 Electrodes High Precision Digital Scale
Change in systolic blood pressure. | Baseline and week 4
  Blood pressure will be measured using the Oklar Blood Pressure Monitors for Home Use Rechargeable Blood Pressure Cuff Wrist Digital BP Machine
Change in lean mass | Baseline and week 4
  Lean mass will be measured using the Runstar Scale for Body Weight and Fat Percentage, 8 Electrodes High Precision Digital Scale
Change in diastolic blood pressure. | Baseline and week 4
  Blood pressure will be measured using the Oklar Blood Pressure Monitors for Home Use Rechargeable Blood Pressure Cuff Wrist Digital BP Machine
WFPB diet acceptability | Post- intervention (day 29)
  At Day 29, participants will complete a Likert-scale survey evaluating the acceptability of the intervention, including satisfaction with meal prep, support sessions, and educational materials. Each item will be rated on a 5-point scale (1 = strongly disagree to 5 = strongly agree). Higher average scores reflect greater acceptability.

SECONDARY OUTCOMES:
Qualitative Assessment of Spousal Influence on Diet Adherence (Exit Interview Coding) | Baseline, post intervention week 4
  Exit interviews will be conducted with a subset of participants in dyads to assess how spousal involvement influenced WFPB diet adherence. Interviews will be transcribed and analyzed thematically. Themes will be identified using qualitative coding methods to evaluate facilitators and barriers related to spousal support. The presence or absence of key support behaviors (e.g., shared cooking, encouragement, resistance) will be documented.
Difference in WFPB Diet Adherence Between Spousal Dyads and Single Individuals | Pre/Post (baseline and 4 weeks)
  Adherence to a whole-food, plant-based (WFPB) diet will be measured using the ACLM Diet Screener at baseline (Day 0) and post-intervention (Day 29), with scores ranging from 0 to 100. Higher scores indicate greater adherence. The change in diet screener scores will be compared between participants enrolled as part of a spousal dyad and those enrolled as individuals to assess whether spousal participation is associated with greater adherence to the WFPB diet.

CONTACTS AND LOCATIONS:
Overall Officials: Brandi White, PhD, Study Chair — University of Kentucky
Locations (1):
- University of Kentucky, Lexington, Kentucky, United States

IPD SHARING:
Plan to Share IPD: No